CLINICAL TRIAL: NCT03429517
Title: Evaluation of Triglycerides and HDL-C Levels in Patients With Acute Coronary Syndrome and Normal LDL-C Level
Brief Title: Levels of Triglycerides and HDL-C in ACS Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Michael Abdo, Principal investigator, Assiut University
Other Study IDs: TGHCACS
Record Dates: First submitted 2018-02-06; First posted 2018-02-12 (Actual); Last update posted 2019-05-10 (Actual); Status verified 2019-05

CONDITIONS: Dyslipidemia Associated With Acute Coronary Syndrome
Keywords: HDL-C; Triglycerides; Non HDL-C and Acute coronary syndrome
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients: ACS Lipogram
  Interventions: Diagnostic Test: Lipogram
- Controls: Normal LDL-C level Lipogram
  Interventions: Diagnostic Test: Lipogram

INTERVENTIONS:
Diagnostic Test: Lipogram — liporgram samples

SUMMARY:
Background Changes in high-density lipoprotein cholesterol and triglyceride levels have been linked to residual cardiovascular risk, whereas non-high density lipoprotein levels have been shown to be more predictive of cardiovascular risk than are low-density lipoprotein cholesterol levels. We aimed to investigate the impact of high density lipoproteins, triglyceride, and non-high density lipoproteins levels on acute coronary syndrome risk with on-target low density lipoproteins levels.

DETAILED DESCRIPTION:
Dyslipidemia: A disorder of lipoprotein metabolism, including lipoprotein overproduction or deficiency. Dyslipidemias may be manifested by elevation of the total cholesterol, the "bad" low-density lipoprotein (LDL) cholesterol and the triglyceride concentrations, and a decrease in the "good" high-density lipoprotein (HDL) cholesterol concentration in the blood. LDL cholesterol is considered the "bad" type of cholesterol. That's because it can build up and form clumps or plaques in the walls of your arteries. Too much plaque in the arteries of your heart can cause a heart attack. HDL is the "good" cholesterol because it helps remove LDL from blood.

HDLs exert multiple anti-atherogenic (inhibition of monocyte adhesion, inhibition of LDL-cholesterol oxidation and MCP-1 expression) and anti-thrombotic effects (decrease platelet aggregability) that together are consistent with a marked reduction in the risk of a morbid cardiovascular event.

Triglycerides come from the calories you eat but don't burn right away, they stored in fat cells and released as energy when you need them Elevated triglycerides have inflammatory (increase the expression of proinflammatory genes (eg, interleukin-6, intercellular adhesion molecule-1, vascular cell adhesion molecule-1, and monocyte chemotactic protein-1), atherogenic (promote proatherogenic responses in macrophages and endothelial cells, possess unique constituents that may contribute to atherogenicity and their by-product (ie, RLPs) may lead to foam cell formation) and thrombotic(increase the expression of coagulation factors or leukocyte adhesion molecules), they also may interfere with the ability of HDL to suppress inflammatory responses in cultured endothelial cells and the capacity of apo AI or HDL to promote sterol efflux from monocytes or macrophages.

The relationship between atherogenic dyslipidemia and cardiovascular risk has been known for decades; however, to date, therapeutic approaches have primarily focused on the lowering of the apoB-containing low-density lipoprotein (LDL) particles. Statin therapy was proven to be effective in the reduction of cardiovascular risk and progression of atherosclerosis. Treatment guidelines are targeted at reaching very low LDL-C levels in high-risk patient groups; however, some studies indicated a residual risk for further cardiovascular events in patients achieving target LDL-C levels with statin therapy.

One potential impediment limiting further reduction in CHD events despite low on-treatment LDL-C is residual elevation in serum triglyceride (TG) levels . Historically, elevated TG has predicted CHD events in univariate analysis, only to weaken after adjustment for other covariates, including plasma glucose and high-density lipoprotein cholesterol (HDL-C), to which it is strongly and inversely correlated Yet, even after adjustment for HDL-C, detailed evaluation of population-based prospective studies has disclosed an independent effect of TG on CHD events . Coupled with the knowledge that combined hyperlipidemia (i.e., elevated LDL-C and TG) promotes CHD to a significantly greater extent than either high LDL-C or TG alone .

Prospective cohort studies, as well as randomized controlled trials of antidyslipidemic therapies, support a powerful inverse correlation between circulating HDL-C levels and coronary risk among patients with elevated, normal, or low low-density lipoprotein cholesterol (LDL-C)

ELIGIBILITY:
Inclusion Criteria:

* ACS
* Normal LDL-C
* Not on statin therapy

Exclusion Criteria:

* Liver disease
* Drug abuse
* End stage renal disease
* Nephrotic syndrome
* Drug abuse

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with a first or subsequent ACS will be enrolled in our study, who are admitted to CCU of Assiut university hospital and Sohag cardiac & digestive system center, more over patients should have LDL-C level below 130mg/dl and lipid samples should be obtained within 4 days of admission. They also should receive treatment according to ACS guidelines.
  Patients and control group data will be collected during a year .
  Patients will be subjected to:
  -Full History taking including : History of chest pain or dysnpea History of renal or liver diseases History of drug abuse History of diabetes and hypertension Family history of cardiovascular diseases and dyslipidemia Assessment of risk factors: smoking, alcohol intake, physical inactivity and poor quality diet.
  Patient Examination :
  Full general and cardiac examination including :
  Xanthelasma Body mass index Waist circumference
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2018-06-01 (Actual); Primary Completion 2019-06-01 (Estimated); Study Completion 2020-06-01 (Estimated)

PRIMARY OUTCOMES:
Decrease ACS events | 1 year
  ACS and Dyslipidemia

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Assiut university hospital, Asyut
  - Sohag Cardiac and Digestive System Center, Sohag

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Baigent C, Keech A, Kearney PM, Blackwell L, Buck G, Pollicino C, Kirby A, Sourjina T, Peto R, Collins R, Simes R; Cholesterol Treatment Trialists' (CTT) Collaborators. Efficacy and safety of cholesterol-lowering treatment: prospective meta-analysis of data from 90,056 participants in 14 randomised trials of statins. Lancet. 2005 Oct 8;366(9493):1267-78. doi: 10.1016/S0140-6736(05)67394-1. Epub 2005 Sep 27. PMID 16214597